CLINICAL TRIAL: NCT02140281
Title: A Phase 1, Single-center, Randomized, 2-Way Cross-over, Open-label Study to Evaluate the Effect of Oral Repeated Doses of AZD1722 on the Pharmacokinetics of Oral Cefadroxil in Healthy Volunteers
Brief Title: To Assess the Effect of AZD1722 on the Pharmacokinetics of Cefadroxil in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5613C00004
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers
Keywords: Phase I, Healthy Volunteers
MeSH Terms: interventions — Cefadroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Treatment A/B) (Experimental): Subjects will be randomised to receive Treatment A in Period 1 followed by Treatment B in period 2
  Interventions: Drug: Treatment A (cefadroxil alone); Drug: Treatment B - AZD1722 followed by cefadroxil
- Sequence 2 (Treatment B/A) (Experimental): Subjects will be randomised to receive Treatment B in Period 1 followed by Treatment A in period 2
  Interventions: Drug: Treatment A (cefadroxil alone); Drug: Treatment B - AZD1722 followed by cefadroxil

INTERVENTIONS:
Drug: Treatment A (cefadroxil alone) — A single 500 mg oral dose of cefadroxil will be given on the morning of Day 1
Drug: Treatment B - AZD1722 followed by cefadroxil — 15mg oral dose of AZD1722 will be given twice daily from Day 1 to Day 4 followed on the morning of Day 5 by a single dose of 15 mg AZD1722 taken together with a single 500mg dose of cefadroxil

SUMMARY:
A study to evaluate the effect of repeated oral doses of AZD1722 on the pharmacokinetics of Cefadroxil

DETAILED DESCRIPTION:
A Phase 1, Single-center, Randomized, 2-Way Cross-over, Open-label Study to Evaluate the Effect of Oral Repeated Doses of AZD1722 on the Pharmacokinetics of Oral Cefadroxil in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:- 1. Healthy male and female volunteers aged ≥18 years to ≤50 years (inclusive) with suitable veins for cannulation or repeated venepuncture 2. Females could be of non-childbearing potential and child bearing potential Females of non-child bearing potential should be Post-menopausal, documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation. Females of childbearing potential must have a negative pregnancy test at screening and must not be lactating, using one of the following effective methods to avoid pregnancy during the treatment periods, must have an established use of oral, injected, or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system, use a barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal. Male healthy volunteers with a partner of childbearing potential must agree to avoid fathering a child, and refrain from donating sperm, from the first day of dosing until at least 3 months after last dose of investigational product, and therefore be either sterile (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate) or agree to use, one of the following approved methods of contraception: a male condom with spermicide; a sterile sexual partner or use by female sexual partner of an acceptable form of effective contraception (see above) 3. Have a body mass index (BMI) ≥18 and ≤30 kg/m2 and weigh at least 50 kg and no more than 100 kg Exclusion Criteria: 1.History of any clinically significant disease or disorder which, in the opinion of the principal investigator, may either put the healthy volunteer at risk because of participation in the study, or influence the results or the healthy volunteer's ability to participate in the study. 2.History or presence of GI, hepatic or renal disease including GI surgery other than appendectomy or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs. 3.Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the investigational product. 3 History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the principal investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD1722 or cefadroxil. 4. Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within at least 30 days of the first administration of investigational product in this study. 5. Loose stools for ≥2 days in the past 7 days before investigational product administration. Use of medications that are known to affect stool consistency and/or GI motility, including fibre supplements, anti diarrheals, prokinetic drugs, enemas, probiotic medications or supplements; or salt or electrolyte supplements containing sodium, potassium, chloride, or bicarbonate formulations during the past 7 days before randomization

Ages: 18 Days to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of cefadroxil when administered after AZD1722 by assessment of area under the concentration-time curve (AUC) and maximal plasma concentration (Cmax) of cefadroxil | Blood sampling for cefadroxil: Predose, 0.5 hour, 1, 1.5, 2, 2.5, 4, 6, 8, 10, and 12 hours postdose on Day 1 in Treatment A and on Day 5 in Treatment B
  Change in plasma area under the concentration-time curve (AUC) and maximal plasma concentration (Cmax) of cefadroxil after AZD1722 administration.

SECONDARY OUTCOMES:
To evaluate the plasma concentrations of AZD1722 | Blood sampling for AZD1722: Predose, 1, 2, and 4 hours postdose, on Day 5 (Treatment B)
  To evaluate plasma concentrations of AZD1722 to be measured (no PK parameters derived)
To evaluate the pharmacodynamic outcomes of AZD1722 by the assessment of how AZD1722 effects stool consistency and frequency | Stool frequency and stool consistency will be measured daily (24-hour period intervals) on Day -1 through Day 1 (Treatment A) and Day 1 through Day 5 (Treatment B)
  Pharmacodynamic outcome of the effect on stool consistency and frequency

OTHER OUTCOMES:
To evaluate the safety profile when cefadroxil is administered after AZD1722 in terms of adverse events, vital signs, electrocardiogram, hematology, clinical chemistry, urinalysis and physical examination | Safety assessments performed through the screening period (Day -28) to 10 days after the last dose in Period 2
  Description of the safety profile in terms of adverse events, vital signs, electrocardiogram, hematology, clinical chemistry, urinalysis and physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor - Lisbon, MD, Principal Investigator — Quintiles, Overland Park, Kansas
Locations (1):
- Research Site, Overland Park, Kansas, United States